CLINICAL TRIAL: NCT03827356
Title: "Comparison Between Two Programs of Inspiratory Muscle Training, Low Resistance vs High Resistance, in Institutionalized Older Women"
Brief Title: "Inspiratory Muscle Training in Older Women"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, CARLOS MARTIN SANCHEZ, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27112018
Record Dates: First submitted 2019-01-28; First posted 2019-02-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Respiratory Insufficiency
Keywords: REHABILITATION; RESPIRATION; BREATHING EXERCISE; FATIGUE; PHYSICAL CAPACITY
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration; Fatigue

STUDY DESIGN:
Intervention Model Description: Patients are assigned randomly to the 2 working groups, each patient only receives one of the two protocols.
Who Masked: Investigator
Masking Description: The principal investigator doesn´t know the group of the patients until the study ends
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "High intensity group" (Experimental): Intervention is administrated with an inspiratory muscle trainer (IMT). High intensity group: 15 cycles, 1 minute each one, 40% MIP with IMT. 1 minute to rest between cycles.
  Interventions: Device: Inspiratory muscle trainer (IMT)
- "Low intensity group" (Active Comparator): Intervention is administrated with an inspiratory muscle trainer (IMT). Low intensity group: 15 cycles, 1 minute each one, 20% MIP with IMT. 1 minute to rest between cycles.
  Interventions: Device: Inspiratory muscle trainer (IMT)

INTERVENTIONS:
Device: Inspiratory muscle trainer (IMT) — The device incorporate a unidirectional valve independent of flow to guarantee constant resistance and included a specific pressure setting (in cm H2O).

SUMMARY:
Objective: To evaluate the effectiveness of two protocols of inspiratory muscle training (IMT) in older women to improve respiratory strength, spirometric parameters and dyspnea. Low-intensity vs high-intensity resistance training programs. Evaluations: Determination of the maximum inspiratory pressure (MIP) and the maximum expiratory pressure (MEP); spirometry - maximum voluntary ventilation (MVV), peak expiratory flow (PEF), tidal volume (TV); functional capacity measured with 6 minute walk test; dyspnea using the Borg scale and clinical evaluations. The participants will be evaluated at the beginning and end of the intervention period. Intervention: There are two groups of patients, one works with low loads (20% MIP) and another with high loads (40% MIP). They train 5 days/week 15 cycles lasting 1 minute. There is a rest of 1 minute between each cycle.

DETAILED DESCRIPTION:
Participants:

Institutionalized women will be recruited to participate in an 8-week randomized trial.

All patients will be asked to carry out the 5-day weekly program, and a recording sheet will be provided to each participant so they will can record the time of each daily respiratory training session. All participants signed an informed consent form.

The patients will be assigned to the two groups randomly. The main researcher doesn´t meet any of the participants until the initial assessment will be carried out.

Evaluation:

The participants are evaluated at the beginning and end of the intervention period.

The evaluation of MIP and MEP is performed using a pressure transducer, Elka 15, which obtains each measurement in millibar and converts it into the reference unit of centimeter of water (cm H2O) (1 mbar = 1.01973 cm H2O .), following the rules of the American thoracic society/European respiratory society (ATS / ERS). The procedure will be repeated until 3 values were obtained with a difference of less than 5%, and the highest value will be used for the analysis. The MIP of the intervention group will be assessed every 2 weeks to set the IMT workload.

Lung volumes are assessed using a spirometer (model: datospir touch) with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules will be followed [19], and the highest value of three correct measurements will be chosen. Data is collected for the following parameters: maximum voluntary ventilation (MVV), forced expiratory volume in the first second (FEV1), peak expiratory flow (PEF), mean expiratory flow (FEF25-75), vital capacity (VC), tidal volume (TV) and forced vital capacity (FVC).

Dyspnea will be measured using the modified Borg scale [20]. Functional capacity will be measured with 6 minute walk test. All evaluations will be done in the corresponding center, during the same time slot and by the same examiner for both groups.

Intervention:

"High-intensity group". The device incorporates a unidirectional valve independent of flow to guarantee constant resistance and includes a specific pressure setting (in cm H2O).

The intensity of the device will be 40% of MIP. The protocol includes 15 cycles lasting 1 minute, twice a day: one in the morning and one in the afternoon. The participants rest for 1 minute between each cycle. In total, the protocol includes 30 minutes of daily respiratory training. The patients will be instructed to inhale with enough force to reach the opening of the valve.

"Low-intensity group".The device incorporates a unidirectional valve independent of flow to guarantee constant resistance and includes a specific pressure setting (in cm H2O).

The intensity of the device will be 20% of MIP. The protocol includes 15 cycles lasting 1 minute, twice a day: one in the morning and one in the afternoon. The participants rest for 1 minute between each cycle. In total, the protocol includes 30 minutes of daily respiratory training. The patients will be instructed to inhale with enough force to reach the opening of the valve.

ELIGIBILITY:
Inclusion criteria:

* Women
* Older 65 years
* Barthel > 60
* Understand the objectives and be able to complete questionaires

Exclusion criteria:

* Respiratory pathology during the 4 weeks prior the start of the study
* Any complication that may impeded the performance of the evaluation tests or breathing techniques

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Female
Enrollment: 26 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (MIP) | 2 minutes
  The evaluation is performed using a pressure transducer, Elka 15, which obtainer each measurement in millibar and converted it into the reference unit of centimeter of water (cm H2O) (1 mbar = 1.01973 cm H2O), following the rules of the American Thoracic Society/European Respiratory Society (ATS / ERS). The procedure was repeated until 3 values were obtained with a difference of less than 5%, and the highest value was used for the analysis. The MIP of the intervention group was assessed every 2 weeks to set the IMT workload.
Maximal expiratory pressure (MEP) | 2 minutes
  The evaluation is performed using a pressure transducer, Elka 15. It is evaluated at the beginning and at the end of the interventional phase.

SECONDARY OUTCOMES:
Maximum voluntary ventilation (MVV) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: Liter (L)/Minute (min)
Forced expiratory volume in the first second (FEV1) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: L
Peak expiratory flow (PEF) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: L/second (seg)
Mean expiratory flow (FEF25-75) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure L/seg
Vital capacity (VC) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: L
Tidal volume (VT) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: L
Forced vital capacity (FVC) | 1 minute
  Spirometer with a turbine transducer with a maximum flow of 16 l/s and a maximum volume of 10 l. The ATS/ERS rules were followed [19], and the highest value of three correct measurements was chosen. Measure: L
Functional capacity | 6 minutes
  The 6 minutes walk test provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
Dyspnea | 1 minute
  Modified Borg scale. It is a numerical scale graduated between 0 and 10, where 0 is the minimum or without dyspnea and 10 is the maximum or extreme dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: ANA MARIA MARTIN-NOGUERAS, DR, Study Chair — University of Salamanca
Locations (1):
- Carlos Martin Sanchez, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No